CLINICAL TRIAL: NCT01754441
Title: Mechanisms of Cell Death in Spinal Muscular Atrophy
Status: Completed | Type: Observational
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Principal Investigator, Matthew E. R. Butchbach, Ph.D., Research Scientist, Nemours Children's Clinic
Other Study IDs: 82008
Record Dates: First submitted 2012-12-13; First posted 2012-12-21 (Estimated); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Spinal Muscular Atrophy
Keywords: Spinal Muscular Atrophy; SMA; Motor Neuron Abnormalities
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Skin biopsy specimens
Oversight: Data Monitoring Committee: No

SUMMARY:
Spinal muscular atrophy is a genetically based disease that affects motor neurons in the spinal cord and leads to muscle wasting and weakness. The gene found to be responsible for the underlying disease is called the SMN or survival motor neuron gene. Individuals with SMA are either missing a copy of the gene or have a mutation in the gene. Although the gene has been identified, how it actually causes the motor neurons to die and leads to muscle wasting and weakness is not completely understood. The investigators have found that skin cells from children with SMA tend to be more susceptible to cell death when exposed to cell death inducing agents. In this protocol, The investigators wish to study the mechanisms by which these cells die when exposed to these agents and how this may be related to the gene defect and the disease.

DETAILED DESCRIPTION:
Spinal muscular atrophy (SMA) is a neuromuscular disease characterized by degeneration of motor neurons and progressive muscle atrophy. The disease is one of the most common genetic causes of infant death. The gene responsible for SMA, survival motor neuron (SMN), exists in humans as two nearly identical copies (SMN1 and SMN2). Only deletion or mutation(s) of the telomeric copy of the gene (SMN1) causes the disease. The SMN protein has been known to function in assembly of the RNA splicing complex, however, the mechanism(s) by which SMN-deficiency causes cell death in SMA are not clear. The long-term goal is to understand the mechanism(s) of motor neuron death in SMA and develop a means of prevention. SMN protein has been reported to have some survival promoting functions in cultured cells. Preliminary studies show that skin fibroblasts from SMA patients are more sensitive to certain death promoting stimuli than control fibroblasts. The investigators hypothesize that the SMN protein is directly involved in cell survival and that loss of this survival function of SMA results in motor neuron death in SMA. The investigators will use fibroblasts from SMA patients, fibroblasts from controls without SMA, motor neuron-like cell lines (such as NSC-34) and rodent primary motor neuron cultures as model systems to test our hypothesis. The investigators will determine the effect of expression of SMN protein in regulating cell death of SMA fibroblasts. The investigators will further investigate the role of SMN in neuronal cell survival. Finally, the investigators will determine biological pathway(s) of SMN-mediated cell protection. Results from the proposed studies will provide insight into the mechanism(s) by which SMN protects cells from death and how a decrease in SMN function leads to the SMA phenotype. Ultimately, the obtained information could lead to develop therapeutic strategies for SMA.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SMA confirmed by neurologist

Exclusion Criteria:

* Not seen as a patient at a participating Nemours facility

Max Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: This study will enroll Children with Spinal Muscular Atrophy (SMA)
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2008-05; Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
SMN localization in SMA fibroblasts | up to 2 years
  Established fibroblast lines from SMA patients will be immunolabeled with antibodies directed against SMN and examined for changes in the nuclear localization of SMN in gems.

SECONDARY OUTCOMES:
SMN isoform mRNA levels | up to 2 years
  The levels of full-length SMN and SMNdelta7 (lacking exon 7) mRNA transcripts will be measured using quantitative PCR.
Protein levels of putative SMA phenotypic modifiers | up to 2 years
  The levels of previously identified modifiers of SMA clinical phenotype (i.e. plastin-3 and ZPR-1) will be examined by immunoblot.
cell viability in response to DNA damaging agents | up to 2 years
  The responsiveness of SMA fibroblasts to DNA damaging agents such as camptothecin, etoposide, bleomycin and actinomycin D will be measured using cell viability assays
SMN protein levels | up to 2 years
  SMN protein levels will be measured by immunoblot.
cell viability in response to cell death-inducing agents | up to 2 years
  The responsiveness of SMA fibroblasts to cell death-inducing agents such as staurosporine, tunicamycin and hydrogen peroxide will be examined using cell viability assays.
SMN2 copy number | up to 2 years
  SMN2 copy number will be determined by quantitative PCR of genomic DNA isolated from established fibroblast lines.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew ER Butchbach, Ph.D., Principal Investigator — Nemours Biomedical Research
Locations (2):
- United States (2):
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Nemours Children's Specialty Care, Jacksonville, Jacksonville, Florida

IPD SHARING:
Plan to Share IPD: Undecided
De-identified data will be made available after publication.

REFERENCES:
- [Result] Stabley DL, Harris AW, Holbrook J, Chubbs NJ, Lozo KW, Crawford TO, Swoboda KJ, Funanage VL, Wang W, Mackenzie W, Scavina M, Sol-Church K, Butchbach ME. SMN1 and SMN2 copy numbers in cell lines derived from patients with spinal muscular atrophy as measured by array digital PCR. Mol Genet Genomic Med. 2015 Jul;3(4):248-57. doi: 10.1002/mgg3.141. Epub 2015 Mar 21. PMID 26247043
- [Result] Stabley DL, Holbrook J, Harris AW, Swoboda KJ, Crawford TO, Sol-Church K, Butchbach MER. Establishing a reference dataset for the authentication of spinal muscular atrophy cell lines using STR profiling and digital PCR. Neuromuscul Disord. 2017 May;27(5):439-446. doi: 10.1016/j.nmd.2017.02.002. Epub 2017 Feb 6. PMID 28284873